CLINICAL TRIAL: NCT06216080
Title: Dynamic Full-Field Optical Coherence Tomography for Structural and Microbiological Characterization of Central Venous Catheter-deposited Biofilm in Critically Ill Patients
Acronym: OCT-BIO-CVC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier William Morey - Chalon sur Saône (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OCT-BIO-CVC
Record Dates: First submitted 2024-01-01; First posted 2024-01-22 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-01

CONDITIONS: Healthcare Associated Infection; Critically Ill; Central Venous Catheter Associated Bloodstream Infection
MeSH Terms: conditions — Cross Infection; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OCT-BIO-CVC cohort: Adult critically ill patients (> 18 years of age) exposed to central venous catheter for at least two calendar days
  Interventions: Other: D-FF-OCT analysis of CVC

INTERVENTIONS:
Other: D-FF-OCT analysis of CVC — Dynamic full-field optical coherence tomography analysis of central venous catheter sections to better apprehend strucural characterization of central venous catheter-deposited biofilm

SUMMARY:
29.3% of bacteremias in intensive care units (ICU) are linked to vascular devices, with a significant proportion related to central venous catheters, and an influence on both morbility and mortality.

It is now accepted that microbiological biofilm plays a key role on both bacterial and fungal development on inner surface of vascular devices but there is yet a lack of clinical relevant data documenting a causal relation between biofilm formation and bacteremias.

We assume that a more precise characterization of central venous catheter-deposited biofilm could help us better understand invasive medical device-related healthcare infections in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient or relative informed of the study and having declared their nonobjection
* Patient over 18 years of age
* Patient exposed to central venous catheter for at least two calendar days

Exclusion Criteria:

* Patient unable to declare their nonobjection
* Patient whose central venous catheter collection is impossible
* Patient admitted in ICU with a central venous catheter already in place

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years of age having declared their nonobjection and exposed to central venous catheter for at least two calendar days
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
D-FF-OCT-based biofilm structure type | At Day 0, within 24h following catheter removal
  Biofilm structure type (ribbon-shaped or mushroom-shaped), measured with D-FF-OCT

SECONDARY OUTCOMES:
D-FF-OCT-based biofilm thickness | At Day 0, within 24h following catheter removal
  Biofilm thickness, measured with D-FF-OCT
D-FF-OCT-based dynamic signal distribution | At Day 0, within 24h following catheter removal
  Biofilm dynamic signal distribution, measured with D-FF-OCT

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maldiney, Principal Investigator — William Morey General Hospital (Chalon-sur-Saône)
Locations (1):
- William Morey General Hospital (Chalon-sur-Saône), Chalon-sur-Saône, Saône-et-Loire, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perez-Granda MJ, Guembe M, Cruces R, Barrio JM, Bouza E. Assessment of central venous catheter colonization using surveillance culture of withdrawn connectors and insertion site skin. Crit Care. 2016 Feb 2;20:32. doi: 10.1186/s13054-016-1201-0. PMID 26838274
- [Background] Silva Paes Leme AF, Ferreira AS, Alves FA, de Azevedo BM, de Bretas LP, Farias RE, Oliveira MG, Raposo NR. An effective and biocompatible antibiofilm coating for central venous catheter. Can J Microbiol. 2015 May;61(5):357-65. doi: 10.1139/cjm-2014-0783. Epub 2015 Mar 2. PMID 25826042